CLINICAL TRIAL: NCT06941467
Title: Efficacy of Topical 0.5% Timolol Solution for Healing Lower Extremity Wounds
Brief Title: Topical 0.5% Timolol Solution for Healing Lower Extremity Wounds
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jesse Lewin, Vice Chair of Surgical Operations, System Chief of the Division of Dermatologic & Cosmetic Surgery, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-23-01193
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Wound Healing; Mohs Micrographic Surgery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Timolol (Experimental): Participants in the topical timolol group will be instructed to apply 1-3 drops of topical 0.5% timolol solution daily to the wound.
  Interventions: Drug: Timolol Maleate Solution
- Standard of Care (Active Comparator): Standard of Care - Apply Vaseline and Band-Aid to wound bed daily
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Timolol Maleate Solution — Timolol 0.5% solution. The number of drops delivered will be based on the initial wound size and will remain constant for the duration of the study period or until the wound is fully re-epithelialized which will be determined by the PI either by photo or in person visit.
  Arms: Timolol
Other: Standard of Care — Vaseline
  Arms: Standard of Care

SUMMARY:
Topical timolol, a β2-Adrenergic receptor (B2AR) antagonist, has demonstrated promise in wound healing over the past several years. The majority of the literature has evaluated the use of topical timolol to shorten wound healing time in chronic wounds of non-surgical etiologies. To date, there are no prospective randomized clinical trials evaluating the role of topical timolol for shortening wound healing time in acute open surgical wounds.

Therefore, the purpose of this study is to determine whether or not topical timolol solution decreases time to wound healing in patients with defects after Mohs Micrographic Surgery (MMS) that cannot be closed with sutures and are left to heal by second intent. The research team also will look to determine if there is a difference in cosmesis of wounds treated with topical timolol compared to those treated with the standard of care. The present study will primarily focus on wounds in the distal lower extremity as these are most commonly left to heal by secondary intent

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo MMS at 234 East 85th St for a skin cancer that is deemed Mohs
* Appropriate by the Mohs surgery appropriate use criteria
* Have an open surgical wound < 4 cm and > 0.5 cm
* Be ≥18 years of age
* English-speaking
* Provide a signed and dated informed consent form
* State willingness to comply with all study procedures

Exclusion Criteria:

* Age less than 18 years of age
* Open surgical wound > 4 cm
* If tumor clearance cannot be achieved with MMS
* Pregnant women
* Breastfeeding women
* Patients who are taking oral beta-blockers (ie oral timolol, metoprolol, carvedilol, propranolol, atenolol)
* Patients who are currently taking any of the following medications: clonidine, digoxin, methyldopa, quinidine, fluoxetine and paroxetine, bupropion
* Patient currently taking a calcium channel blocker AND has pre-existing heart failure as defined by a reduced ejection fraction
* Patients with pre-existing hypotension
* Pre-existing diagnosis of sinus bradycardia
* Pre-existing diagnosis of second or third degree atrioventricular block
* Congestive heart failure
* Pre-existing diagnosis of severe asthma
* Pre-existing diagnosis of chronic obstructive pulmonary disease
* Any known hypersensitivity to 0.5% timolol solution
* Patients who have a wound where primary closure is feasible and desired by the patient
* Defect size <0.5 cm
* Prior sensitivity or known allergy to timolol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Wound surface area healing (skin reepithelialization) | 2 weeks, 4 weeks, 6 weeks, 12 weeks
  The wound surface area healing (skin reepithelialization) in open post-surgical lower extremity wounds will be measured using a ruler.

SECONDARY OUTCOMES:
Percentage change in surgical wound size | 2 weeks, 4 weeks, 6 weeks, 12 weeks
  Percentage change in surgical wound size
Modified Manchester Scar Scale (MMSS) | 2 weeks, 4 weeks, 6 weeks, 12 weeks
  The Modified Manchester Scar Scale (MMSS) is a clinical tool used to evaluate the appearance and characteristics of scars. The MMSS assess four key aspects of the scar:
  * Color (compared to surrounding skin): Rated 1-4
    * Perfect match (1) to gross mismatch (4)
  * Matte vs. Shine: Rated 1-2
    * Matte appearance (1)
    * Shiny appearance (2)
  * Contour: Rated 1-3
    * Flush with surrounding skin (1)
    * Slightly proud/indented (2)
    * Hypertrophic (3)
  * Distortion: Rated 1-4
    * No distortion (1 point) to severe distortion (4 points)
  The total score ranges from 4 to 13, with higher scores indicating a more noticeable or problematic scar.
The Pain, Enjoyment of Life and General Activity scale (PEG) | 2 weeks, 4 weeks, 6 weeks, 12 weeks
  The PEG, a Three-item Scale Assessing Pain Intensity and Interference Pain is is a 3-item questionnaire that measures pain intensity and pain-related functional interference with open wounds on the lower leg. The assessment includes three domains: average pain intensity (0-10), pain interference with enjoyment of life (0-10), and pain interference with general activity (0-10). The total score ranges from 0-30, with higher scores indicating greater pain intensity and greater pain-related functional interference.
Wound Quality of Life Questionnaire (Wound-QOL) | 2 weeks, 4 weeks, 6 weeks, 12 weeks
  The Wound-QoL is a17-item questionnaire assesses how patients feel about their open wound its impact on their quality of life. The assessment evaluates multiple dimensions of wound-related quality of life, including physical symptoms (items 1-3), functional limitations (items 4, 11-15), psychological well-being (items 6-10), and burden of care (items 5, 16-17). Each item is scored on a 5-point scale from "Not at all" (0) to "Very much" (4). The total score ranges from 0-68, with higher scores indicating lower wound quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Lewin, MD, Principal Investigator — Primary Investigator
Locations (1):
- Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in ISMMS data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (to be determined).